CLINICAL TRIAL: NCT00158873
Title: A Centre-Randomized, Open-Label, Cross-Over Study to Compare the Pharmaco-Economic Consequences of an Ultiva (Remifentanil Hydrochloride) Based Regimen With Conventional Sedative Based Regimens in ICU Subjects Requiring Short-Term Mechanical Ventilation With Analgesia and Sedation
Brief Title: Pharmaco-Economic Study Of Ultiva In Intensive Care Unit(ICU)Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 101653
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Sedation
Keywords: ICU mechanical ventilation analgesia sedation
MeSH Terms: interventions — Midazolam; Lorazepam; Fentanyl; Morphine; Remifentanil; Propofol

INTERVENTIONS:
Drug: midazolam
Drug: lorazepam
Drug: fentanyl
Drug: morphine
Drug: remifentanil
Drug: propofol
  Other Names: midazolam; lorazepam; fentanyl; morphine; remifentanil

SUMMARY:
The study will evaluate the pharmaco-economic consequences of the use of a remifentanil based regimen compared with a conventional sedative based regimen in terms of duration of mechanical ventilation, length of stay in ICU, difference in extubation time and use of concomitant sedative agents.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with an expected duration of mechanical ventilation for 2 to 3 days and requiring analgesia and sedation.

Exclusion criteria:

* ICU patients resuscitated in the previous 24 hours, neurotrauma or expecting major surgery, not likely to survive of with limit care status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224
Dates: Start 2004-09

PRIMARY OUTCOMES:
Health Outcome: Duration of time on mechanical ventilation

SECONDARY OUTCOMES:
Health Outcome: length of stay in ICU, in hospital, requirement of opioid and sedative agents, duration of extubation process. Safety: haemodynamics and adverse events. Efficacy: sedation and pain scores

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (15):
- Netherlands (15):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Apeldoorn
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Haarlem
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tiel
  - GSK Investigational Site, Venlo
  - GSK Investigational Site, Zwolle

REFERENCES:
- [Derived] Al MJ, Hakkaart L, Tan SS, Bakker J. Cost-consequence analysis of remifentanil-based analgo-sedation vs. conventional analgesia and sedation for patients on mechanical ventilation in the Netherlands. Crit Care. 2010;14(6):R195. doi: 10.1186/cc9313. Epub 2010 Nov 1. PMID 21040558